CLINICAL TRIAL: NCT04444947
Title: Influencing Factors in Patients With Colorectal and Gastric a Retrospective Study
Brief Title: Influencing Factors in Patients With Colorectal and Gastric Polyps a Retrospective Study
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-SR-340
Record Dates: First submitted 2020-06-11; First posted 2020-06-24 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Polyp, Colonic
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The identification of risk factors of colorectal/gastric polyp is more helpful for preventing colorectal cancer. And modifiable factors (such as high-fat diet, abnormal blood lipid, smoking, lack of exercise, obesity), and unmodifiable factors (including age, gender, race, familial adenomas, genetic)) can affect the risk of polyps. Thus early studying risk factors are the key to improving prognosis. what's more, early detection and timely treatment have important clinical significance for preventing and reducing the occurrence of gastrointestinal cancer.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most common cancer in the world. what's more, CRC is therefore an important public health concern in China due to its rising incidence and prevalence, in addition to the burden of disease. There is robust evidence indicating that early detection by screening and removal of cancer precursor lesions offers an effective method of reducing colorectal cancer morbidity and mortality. Studies have shown that colorectal polyps are considered to be related to colorectal cancer, especially adenoma .The primary aim of this study was to identify high risk features of multiple polyps based on size, location and histological type. Patient age and gender were also characterized on the basis of a contingency analysis of a large series of Chinese patients with colorectal polyps. These data provide important information on risk factors associated with multiple polyps, which will serve as evidence for an individualized approach to colonoscopy screening guidelines in China.

Similarly, recent years, with the widespread use of gastroscopy, people's health awareness and lifestyle changes, more and more people have performed gastroscopy, so a large number of patients with gastric polyps can be found in the clinic. Gastric polyps are raised lesions that originate in the mucosal layer or submucosa and protrude into the stomach cavity. According to their pathological characteristics, they can be divided into two categories: mucosal layer and non-mucosal layer.Gastric polyps originating from mucosal layers, represented by natural, fundus glandular and adenomatous polyps, are the most common in clinical practice, while non-mucosal polyps including gastric stromal tumors and inflammatory fibrous polyps are more common in clinical practice. Although the incidence of gastric polyps is far less than that of intestinal polyps, some pathological types, especially adenomatous polyps, have obvious malignant potential and are recognized as precancerous lesions .

Therefore, we retrospectively analyzed the records of patients with gastrointestinal polyps in our hospital in the past years, and provided epidemiological data to study the factors in polyps.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent colonoscopies

Exclusion Criteria:

* (1) Patients with Crohn's disease, inflammatory bowel disease, and colorectal cancer; (2) Patients with ulcerative bowel disease, and intestinal tuberculosis; (3) Patients with history of familial polyposis; (4) All patients without complete endoscopic reports and complete demographics records.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: A total of 43,104, patients (n=21939) with polyps and patients without polyps (n=21165) is included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 64889 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Influencing factors in patients with colorectal polyps: a retrospective study | JUNE 30,2020
  risk factors

CONTACTS AND LOCATIONS:
Overall Officials: yue WANG, master, Principal Investigator — the Human Ethics Committee of Jiangsu Provincial People's Hospital
Locations (1):
- Jiangsu Provincial People's Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Han X, Qian W, Liu Y, Zheng T, Su XJ, Zhang PP, Chen Y, Hu LH, Li ZS. Effects of age, sex and pathological type on the risk of multiple polyps: A Chinese teaching hospital study. J Dig Dis. 2020 Sep;21(9):505-511. doi: 10.1111/1751-2980.12863. PMID 32279448
- [Result] Song M, Emilsson L, Bozorg SR, Nguyen LH, Joshi AD, Staller K, Nayor J, Chan AT, Ludvigsson JF. Risk of colorectal cancer incidence and mortality after polypectomy: a Swedish record-linkage study. Lancet Gastroenterol Hepatol. 2020 Jun;5(6):537-547. doi: 10.1016/S2468-1253(20)30009-1. Epub 2020 Mar 17. PMID 32192628
- [Result] Mariotto AB, Yabroff KR, Shao Y, Feuer EJ, Brown ML. Projections of the cost of cancer care in the United States: 2010-2020. J Natl Cancer Inst. 2011 Jan 19;103(2):117-28. doi: 10.1093/jnci/djq495. Epub 2011 Jan 12. PMID 21228314
- [Result] Oines M, Helsingen LM, Bretthauer M, Emilsson L. Epidemiology and risk factors of colorectal polyps. Best Pract Res Clin Gastroenterol. 2017 Aug;31(4):419-424. doi: 10.1016/j.bpg.2017.06.004. Epub 2017 Jun 28. PMID 28842051